CLINICAL TRIAL: NCT06482515
Title: Take the Reins: The Effects of Nutrient Timing on Cancer-related Fatigue Among Blood Cancer Survivors (2458GCCC)
Brief Title: Take the Reins: The Effects of Nutrient Timing on Cancer-related Fatigue
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Amber Kleckner, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00110284
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms; Blood Cancer; Fatigue; Diet Habit; Survivorship; Fasting, Intermittent
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Fatigue; Feeding Behavior; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Time-restricted eating (Experimental)
  Interventions: Behavioral: Time-restricted eating; Behavioral: Nutrition counseling
- Time-unrestricted eating (Active Comparator)
  Interventions: Behavioral: Nutrition counseling

INTERVENTIONS:
Behavioral: Time-restricted eating — Participants will be asked to eat all their food in a self-selected 10-hour eating window every day.
  Arms: Time-restricted eating
Behavioral: Nutrition counseling — Participants will meet with a nutritionist to discuss their dietary habits and how they compare to the American Cancer Society nutrition guidelines.

SUMMARY:
Cancer-related fatigue affects at least 30-90% of patients with cancer, depending on the type of cancer and their treatment(s) (e.g., chemotherapy, radiation). It is not relieved by sleep or rest, and it sometimes can persist for years after a person's cancer was treated. The fatigue can be so bad that people cannot return to work, hobbies, family roles, or other daily activities, thereby greatly reducing quality of life. The causes of this fatigue are unknown, and we currently do not have anything that can reliably prevent or cure the fatigue. However, there are recent data suggesting that circadian rhythm, or a person's internal body clock, may be disrupted by the cancer experience and contribute to fatigue. Food intake is an external cue that can entrain circadian rhythm. We recently showed that cancer survivors are willing and able to eat all their food within a 10-hour eating window-a practice called time-restricted eating. Herein, we are testing time-restricted eating against a control group (matched for time-, attention, and expectancy) to see if time-restricted eating can indeed alleviate cancer-related fatigue. All participants will be asked to use the myCircadianClock smartphone app to log their food intake and weekly body weight measurements. The participants assigned to the time-restricted eating group will be asked to eat all their food in a 10-hour window during the day. People can choose their start time based on their schedule and preferences, but we ask that the window is the same for the whole study (e.g., 7am-5pm,9:30am-7:30pm). Black coffee and unsweetened tea are allowed before the eating window, and water and medicines are allowed at all times. The participants in the control group will meet with a nutritionist to discuss the American Cancer Society nutrition guidelines in cancer survivorship; they will not be restricted to when they can eat. Participants in both groups will give us valuable information regarding how diet is related to the experience of fatigue. The purpose of this study is to test the effects of a 12-week TRE intervention vs. an unrestricted eating pattern on fatigue, the sustainability of the program at 24 weeks, and the effects of TRE on circadian rhythm and sugar metabolism.

ELIGIBILITY:
Inclusion criteria (Participants must…):

* Have a diagnosis of a hematologic neoplasm (e.g., leukemia, lymphoma, multiple myeloma);
* Be at least 2 months post-treatment with chemotherapy, radiation, targeted therapy, chimeric antigen receptor (CAR)-T cell therapy, stem cell transplant, or another therapy (maintenance therapies are okay; steady unchanged treatment for relapsed disease for >2 months and expected to stay on it until progression is okay);
* Have a baseline level of fatigue, as determined by at least one of the following:

  1. Reporting a score of 4 or higher in response to the question, "What was your worst fatigue in the last week, on a scale of 0-10, where 0 is no fatigue and 10 is the worst fatigue?"
  2. In the habit of taking daytime naps,
  3. Have fatigue that interferes with their ability to work, engage in social events, or is more than would be expected from physical exertion,
* Be able to speak and/or read and write in English or Spanish;
* Be at least 18 years old; and
* Be able to provide informed consent.

Exclusion criteria (participants must not…)

* Be underweight, as defined as a body mass index <18.5 kg/m2;
* Already eat all their food within a window that is 10 h or shorter most (6/7) days of the week;
* Be employed in a job where they regularly work away from the home at night (e.g., night shift);
* Have surgery planned during the study duration;
* Have any contraindications to the proposed nutrition intervention as identified by their medical provider, their designee, or the study team (e.g., type 1 diabetes, risk for hypoglycemia, medication requirements, pregnancy, breastfeeding, recent history of an eating disorder);
* Be taking insulin; or
* Be on enteral or parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | baseline, 6 weeks, 12 weeks
  Multidimensional Fatigue Symptom Inventory-Short Form; the total MFSI-SF score ranges from -24 to 96 with a higher score indicating higher levels of fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data files and transcripts will be shared using Dryad (datadryad.org) per guidelines of the data repository, or similar repositories. All de-identified demographic data, clinical record data, and arm allocation from the parent trial will be shared in conjunction with the data to increase the usefulness to other researchers. In addition, the interview guide will be shared in text format (.pdf or .txt). The blank questionnaires will also be shared via the same repository.
Time Frame: Data will be made available when the work is published or the award/support period ends, whichever comes first. Data will be accessible at a minimum of three years post-completion of this award and the parent grant, as required by the federal retention guidelines. We will keep the data available as long as it is useful, which we estimate will be 10-20 years. We hope to have the data accessible indefinitely.